CLINICAL TRIAL: NCT01172041
Title: Investigating the Role of Audiovisual Biofeedback on Image Quality During 4D Anatomic and Functional Imaging
Brief Title: The Role of Audiovisual Biofeedback on Image Quality During 4D Anatomic and Functional Imaging
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: LUN0026; 98393 (Other: Stanford University Alternate IRB Approval Number); SU-05152009-2578 (Other: Stanford University); 10886 (Other: Stanford IRB)
Record Dates: First submitted 2010-07-26; First posted 2010-07-29 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Real time position management system — Device to monitor respiration by using optical monitoring of a marker block placed on the abdomen of the patient.
  Other Names: Varian
Device: LS PET/CT — PET/CT scanner for acquiring CT and PET images (3D and 4D)
  Other Names: GE
Drug: 18-FDG — 15mCi
  Other Names: Fludeoxyglucose (18F); fluorodeoxyglucose (18F)

SUMMARY:
This study will investigate whether audiovisual biofeedback, in which visual and audio cues are used to regulate the patient's breathing, can increase the image quality of 4D CT and 4D PET scans.

ELIGIBILITY:
Inclusion Criteria:

Required for inclusion in this study are:

* Informed consent
* Diagnosis of AJCC Stage I-III lung cancer of any histology to be treated using radiotherapy at Stanford Cancer Center
* Age 18 or greater
* Painfree in supine position
* Karnofsky performance status 50 or greater

The inclusion of educationally disadvantaged, decisionally impaired or homeless people are allowed if informed consent, in the opinion of the consenting investigator (study PI, co-PI or research nurse), is obtained.

Exclusion Criteria:

No

* Pregnant women
* Stanford employees
* Stanford students
* Prisoners will be eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of AJCC Stage I-III lung cancer of any histology to be treated using radiotherapy at Stanford Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Measure the difference in number of artifacts on 4D CT scans using audiovisual biofeedback in comparison to Free breathing. | Day one
  The first, third, fifth seventh and ninth patients accrued to the protocol will have their free breathing studies performed first. The second, fourth, sixth, eighth and tenth patients accrued to the protocol will have their audiovisual (a/v) biofeedback studies performed first.

CONTACTS AND LOCATIONS:
Overall Officials: Bill Loo, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Yang J, Yamamoto T, Pollock S, Berger J, Diehn M, Graves EE, Loo BW Jr, Keall PJ. The impact of audiovisual biofeedback on 4D functional and anatomic imaging: Results of a lung cancer pilot study. Radiother Oncol. 2016 Aug;120(2):267-72. doi: 10.1016/j.radonc.2016.05.016. Epub 2016 May 30. PMID 27256597